CLINICAL TRIAL: NCT06716411
Title: Confirming the Effects of Acupuncture Treatments to Relieve Symptoms of Gulf War Illness
Acronym: CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of California, Berkeley (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Lisa J Taylor-Swanson, Principal Investigator, PhD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TX230133; TX230133 (Other Grant/Funding Number: Department of the Army)
Record Dates: First submitted 2024-08-16; First posted 2024-12-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Persian Gulf Syndrome; Gulf War Syndrome; Multiple Chronic Illnesses; Occupational Diseases; War-Related Injuries; Wounds and Injuries
Keywords: Acupuncture; Gulf War Illness; Complex Medical Illness; Chronic Multisymptom Illness; Veteran
MeSH Terms: conditions — Persian Gulf Syndrome; Multiple Chronic Conditions; Occupational Diseases; War-Related Injuries; Wounds and Injuries | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bi-weekly acupuncture treatment (Experimental): Bi-weekly acupuncture treatment
  Interventions: Device: Acupuncture
- Wait list (Active Comparator): Wait list for 2 months followed by weekly acupuncture for 4 months
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Sterile insertive needles are applied by licensed, experienced practitioners.

SUMMARY:
This unblinded Phase II clinical trial will test the effects of individualized acupuncture treatments offered in extant acupuncture practices in the community; practitioners will have had at least 5 years of experience plus additional training provided by the study. Veterans with diagnosed symptoms of Gulf War Illness will be randomized to either six months of biweekly acupuncture treatments (group 1, n=100) or 2 months of waitlist followed by weekly acupuncture treatments (group 2, n=100). Measurements were taken at baseline, 2, 4 and 6 months. The primary outcome is the SF-36 physical component scale score (SF-36P).

DETAILED DESCRIPTION:
Gulf War Illness (GWI), or chronic multisymptom illness (CMI), is a complex illness characterized by multiple symptoms, including fatigue, sleep and mood disturbances, cognitive dysfunction, and musculoskeletal pain, which are unexplained by physical and laboratory examinations. There is no standard of care treatment for this syndrome at this time. First defined by the Centers for Disease Control and Prevention (CDC) after the first Gulf War, it is commonly seen with a highly individualistic presentation, associated with clusters of symptoms and co-morbid medical diagnoses, including chronic fatigue syndrome, fibromyalgia, irritable bowel syndrome, arthralgia, digestive complaints, and mood-related psychiatric disorders, including depression, posttraumatic stress disorder (PTSD), and other anxiety disorders. It has been shown to be remarkably stable at 5- and 10- year follow-ups. Of the 700,000 service personnel deployed to the Persian Gulf, 100,000 veterans of the first Gulf War (Operation Desert Shield/Storm, years 1990-1991) have presented with medical complaints through clinical and registry programs. GWI is twice as prevalent in deployed veterans, and seen in 15% of non-deployed veterans.

CMI symptoms have been studied in cohorts of veterans in the United Kingdom, Canada, and Australia. The etiology of CMI is still unknown, and hypotheses involving exposures to vaccines, medications, pesticides, chemical munitions, and inhalation of depleted uranium dust and smoke from burning oil fields, have all been investigated inconclusively. Stress plays a likely role in the etiology of other multisymptom illnesses, such as irritable bowel syndrome (IBS), multiple chemical sensitivity and chronic headache. It is likely that veterans of the current war in Iraq and Afghanistan are exposed to similar deployment stressors and will benefit from an investigation of CMI and its treatment.

Acupuncture is an evidence-based, nonpharmacologic treatment commonly used for many symptoms affecting veterans and active military personnel, including pain. Acupuncture has shown efficacy for a variety of painful musculoskeletal disorders, as a treatment for both acute and chronic pain after amputation in military contexts, and in the treatment of related comorbidities such as fatigue, state, trait and situational anxiety, and depression. Acupuncture has shown effectiveness and is used in the Veterans Health Administration (VHA) and covered by Medicare for some conditions.

The L Conboy lab has completed multiple successful acupuncture trials in areas such as Irritable Bowel Syndrome, Carpel Tunnel Syndrome, and pelvic pain. Most recently the study team successfully completed a 3.5-year Congressionally Directed Medical Research Program (CDMRP) randomized controlled trial (RCT) "The Effectiveness of Acupuncture in the Treatment of Gulf War Illness". In that study, veterans chose a trained study acupuncturist in a location convenient to them. These community-based acupuncturists provided personalized acupuncture in a therapeutically informed dose. In the robust sample (n=104), investigators found a clinically and statistically significant improvement in pain after 2 months of treatment. After 6 months of treatment McGill Pain Scale values showed a 6-point improvement (p<=0.001), and the physical component of the SF-36 (SF-36P) showed a 9-point improvement (p<=0.003). Investigators also found statistically and clinically improvements in: the severity of veterans' self-reported main (p<0.01) and secondary (p<0.009) complaints as measured by the patient-centered Measure Your Medical Outcomes Profile (MYMOP) outcome measure, self-reported overall health from the SF-36P (p<0.007), and fatigue (p<0.05) based on the Multidimensional Assessment of Fatigue. Patient satisfaction with care and confidence in treatment was also very high (95% rated satisfied and confident). In addition, investigators found that the theoretically informed dose (2 sessions per week for 6 months) provided more relief for pain and poor function than did the comparison dose of one session per week, and that over 95% of symptom improvement for pain was maintained at 5-year follow up. Acupuncture at a sufficient dose is one of the only treatments found to be effective in improving pain and function in this hard-to-treat population while also addressing other symptoms in the patient's biopsychosocial presentation. Other high-quality science has shown that dosage is important for acupuncture treatment, and that treatment effects can persist long after acupuncture treatment has ended.

While this clinical data is very promising, equally important is furthering the understanding of the mechanisms of Gulf War Illness and successful treatments. Investigators conducted blood biomarker analyses using the collected blood samples from the parent trial, including collaborations with the Boston Biorepository, Recruitment and Integrative Network (BBRAIN) consortium at Boston University. Investigators found a number of interesting contrasts including significantly altered ether lipid metabolism in GWI, and that acyl-carnitine molecules are decreased in GWI, in agreement with previous reports. More recently, in collaboration with anti-aging researchers at Berkeley, investigators have found that acupuncture at the proper dose shifts the protein signature of GWI veteran to resemble a younger state (see below). In order to further elucidate the mechanisms underlying both GWI and successful treatments, the collection of blood biomarkers will be augmented by collection of physiological biomarkers potentially implicated in GWI symptoms.

Autonomic dysregulation has been demonstrated to be common among Veterans with GWI, according to both self-report and objective measures. The 31-item Composite Autonomic Symptom Score (COMPASS-31) scale assesses autonomic dysregulation. COMPASS-31 scores were positively associated with physical function in a GWI population, with gastrointestinal (GI) symptoms as the autonomic subscale most strongly correlated. A pilot study using heart rate variability (HRV) measurement reported parasympathetic activity (PNS) negatively associated with GWI symptoms, while sympathetic nervous system activity (SNS) was positively associated with symptoms. Further, some data suggest that treatment improvements in those with GWI are associated with improvements in autonomic regulation. For example, yoga and breathing techniques have demonstrated in multiple studies in veterans and non-veterans improvements in symptoms associated with GWI, including autonomic symptoms, chronic pain, and irritable bowel syndrome. Exploration of autonomic dysregulation in this study of acupuncture for GWI is thus proposed because acupuncture is associated with decreased autonomic symptoms. A recent meta-analysis concluded that real acupuncture has a superior effect over placebo acupuncture in increasing parasympathetic tone, though this has yet to be studied in GWI.

Gastrointestinal problems and fatigue are also highly prevalent among veterans with GWI. Autonomic dysregulation among veterans with GWI has been studied with respect to gastroparesis as demonstrated by a composite autonomic score of 3.7 in veterans with GI symptoms (vs 1.3 in controls) (p<0.01). Previous work on GWI and HRV on the outcome of fatigue found a significant negative relationship between root mean square of successive differences of beat-to-beat intervals (RMSSD), a measure of PNS activity, and fatigue [r = -.0574]. This is consistent with literature indicating decreased parasympathetic activity to be a characteristic feature of both acute and daily levels of fatigue. Other work on acupuncture and HRV on the outcome of fatigue supports the investigation that acupuncture treatment is associated with decreased autonomic symptoms. Further a recent meta-analysis concluded that real acupuncture has a superior effect over placebo acupuncture in increasing parasympathetic tone, though this has yet to be studied in GWI. One study of acupuncture demonstrated decreased fatigue among patients with Chronic Fatigue Syndrome, and also reported instantaneous changes of HR after acupuncture therapy was administered.

If investigators confirm the previous clinical results, this data set will provide valuable documentation of the clinical, biological, and physiological changes that occur as veterans with GWI move to a healthier state. This will greatly improve current understanding of the Whole Health of GWI veterans, with applications to other clinical modalities and illnesses.

Subjects will be recruited via local advertisements and direct mailing to veterans on the Gulf War Registry, who live in one of the 6 areas identified by the team to have greater density of veterans diagnosed with Gulf War Illness. Through questionnaires, physician assessment, and medical histories, the investigators measured the severity of symptoms before beginning treatment, and after 2, 4 and 6 months of treatment. One group of patients received acupuncture evaluation and treatment twice per week for 6 months. A second group, for comparison purposes, will be monitored on a wait list for 2 months, and will then be offered weekly acupuncture for 4 months. The primary comparison is the difference at 6 months. Based on previous acupuncture research on fatigue, stress, and pain, including the parent study, the investigators expect this length of treatment will be enough for patients to receive significant benefit. The investigators also planed to collect samples of blood from the volunteers that will help identify possible disease mechanisms for the illness and track the effects of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Deployed to the Gulf Theater of operations (as defined by 38 CFR 3.317, includes Iraq, Kuwait, Saudi Arabia, Bahrain, Qatar, the United Arab Emirates, Oman, the Gulf of Aden, the Gulf of Oman, the Persian Gulf, the Arabian Sea, the Red Sea, and the airspace above all of these locations) between August 1990 and the present date
* Have at least 2 of the following symptoms from the 3 CDC clusters of symptom that have lasted for more than 6 months. Each symptom cluster must be characterized as mild-moderate or severe, with at least one symptom in each cluster required to be severe. The clusters are:

A. Fatigability: fatigue 24 hours or more after exertion B. Mood and Cognition: feeling depressed; feeling irritable; difficulty thinking or concentrating; feeling worried, tense, anxious; problems finding words; or problems getting to sleep C. Musculoskeletal: joint pain or muscle pain

Exclusion Criteria:

* Currently enrolled in another clinical trial
* Have another disease that likely could account for the symptoms, as determined by our Medical Monitor
* Severe psychiatric illness (in the last 2 years psychiatric hospitalization, suicidal attempt, alcohol or substance abuse, use of antipsychotic medication) as measured by the Primary Care Evaluation of Mental Disorder (Prime MD).
* Unable to complete the protocol on based on the evaluation of the Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
SF-36P | 6 months
  Ten items addressing physical functioning which are part of a short-form health survey with 36 questions. Scores range between 0 and 100 with higher scores indicating better function.

OTHER OUTCOMES:
Blood Draw | 6 months
  Blood draws will be used to examine levels of selected markers of inflammation, stress, and immune function. The units of measure would be relative to control, baseline or untreated. The following proteins will be evaluated:
  TRAIL-R1 (Tumor necrosis factor-Related Apoptosis-Inducing Ligand Recombinant protein 1); IL-16 (Interleukin 16) TIMP-1 (Tissue Inhibitor of MetalloProteinases-1); IL-15Ra (Interleukin 15 R alpha); CD27 (also known as Tumor necrosis factor receptor superfamily member 7 (TNFRSF7)); APJ (apelin receptor); SMAD5 (mothers against decapentaplegic homolog 5); uPAR (urokinase plasminogen activator surface receptor); FADD (Fas-associated death domain); MFGE8 (Milk fat globule epidermal growth factor 8); ICAM-1 (Intercellular adhesion molecule 1); TNFRSF27 (tumor necrosis factor receptor superfamily member 27); CCL25 (Chemokine ligand 25); TGFbR2 (transforming growth factor beta receptor 2); TLR4 (tool-like receptor 4)
McGill Pain Scale | 6 months
  The McGill Pain scale is perhaps the most recognized and utilized pain measurement device across a range of ailments. This 15-item measure asks participants to describe the quality of their pain using various different descriptors (73). The McGill pain scale is 0-60 range, where the worse the pain the higher the number.
Heart rate variability (HRV) | 6 months (starting two weeks before treatment starts until the end of treatment)
  Signs and symptoms of autonomic dysfunction, including changes in heart rate variability (HRV), have been demonstrated among veterans diagnosed with GWI. Acupuncture has also demonstrated an impact the autonomic nervous system by effecting a shift away from sympathetic dominance and toward parasympathetic dominance. So, we propose to measure HRV parameters as a physiological biomarker of treatment effect. Specifically, the team will gather the following HRV data: heart rate (HR); respiratory rate (RR); standard deviation of normal-to-normal intervals (SDNN); root mean square of successive differences (RMSSD); pNN50 (percentage of consecutive normal sinus intervals that differ by more than 50 milliseconds); VLF (band of rhythms with periods between 25 and 300 s); LF (band of rhythms with periods between 7 and 25 s); any heart failure (HF); LF/HF (ration of low frequency to high frequency); and total power. HRV data will be extracted continuously from Fitbits worn by participants.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of California, Berkeley, Berkeley, California
  - Various, Los Angeles, California
  - Various, Colorado Springs, Colorado
  - Various, Denver, Colorado
  - Various, Tampa, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Various, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Various, Fairfax, Virginia
  - Various, Seattle, Washington